CLINICAL TRIAL: NCT06076031
Title: To Investigate the Effects of Applying Streaming Media on Reducing Pain Medication, Anxiety, and Pain and Related Factors in Patient With Second-degree Burn During Changing Dressing：A Cross-over Randomization Study
Brief Title: Effects of Applying Streaming Media on Reducing Pain in Patient With Second-degree Burn During Changing Dressing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB2023051
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Burns; Pain, Burning; Anxiety
Keywords: second-degree burns; streaming; pain; anxiety; pain medication; dressing change
MeSH Terms: conditions — Burns; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (No Intervention): Analgesic use
- lntervention (Experimental): streaming media (video and audio) use
  Interventions: Behavioral: Streaming Media

INTERVENTIONS:
Behavioral: Streaming Media — The aim of this study is to conduct a cross-over randomized clinical trial to compare the effects of with using streaming media (video and audio) on reducing pain medication use, anxiety, pain intensity, and factors related to pain during dressing changes for second-degree burn patients.
  Arms: lntervention

SUMMARY:
During the acute phase of burn injuries, the focus for patients is primarily on wound pain and infection care. Patients often describe the pain during dressing changes as a sharp, stabbing sensation. Pain is a distressing experience for burn injury patients, affecting both their physical and mental well-being, as well as influencing wound healing. The pain caused by dressing changes is a significant issue that leads to physical and emotional suffering for patients.

DETAILED DESCRIPTION:
Background: During the acute phase of burn injuries, the focus for patients is primarily on wound pain and infection care. In this stage of treatment, frequent dressing changes are necessary, with some wounds requiring daily cleansing to promote healing and prevent infection. Patients often describe the pain during dressing changes as a sharp, stabbing sensation. Pain is a distressing experience for burn injury patients, affecting both their physical and mental well-being, as well as influencing wound healing. The pain caused by dressing changes is a significant issue that leads to physical and emotional suffering for patients.

Objective: The aim of this study is to conduct a cross-over randomized clinical trial to compare the effects of with using streaming media (video and audio) on reducing pain medication use, anxiety, pain intensity, and factors related to pain during dressing changes for second-degree burn patients.

Methods: This study plans to utilize a cross-over randomized clinical trial design with patients from the burn injury ward of a regional teaching hospital in Chiayi. Research instruments include demographic characteristics, disease information, Burn Pain Anxiety Scale, Numerical Pain Scale, and vital signs. Statistical methods will encompass descriptive statistics, independent samples t-test, chi-square test, generalized estimating equations, and multiple linear regression to identify the effectiveness of streaming media usage during dressing changes for second-degree burn patients in reducing pain medication use and anxiety, as well as related factors.

Expected outcomes: It is anticipated that the use of streaming media during dressing changes for second-degree burn patients will lead to reduced pain medication use, anxiety, and related factors. The results of this study can provide evidence for the intervention of using streaming media to alleviate dressing change pain effectively during the care of second-degree burn patients, thereby enhancing the quality of pain care.

ELIGIBILITY:
Inclusion Criteria:

* Must stay in the burn ward for 2 days
* Have clear consciousness
* Aged 20 years old (inclusive) and above superior
* Patients with superficial 2 degree burns accounting for 10% of the body surface area or deep 2 degree burns accounting for 5% of the body surface area were diagnosed by physicians
* Can communicate in Chinese and Taiwanese and agree to participate in this study

Exclusion Criteria:

* Mental disease.
* Cognitive impairment.
* Visual and hearing impairment.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) : 0 means no pain, and 10 means very painful. | one year
  1. The intensity of pain 30 minutes before the dressing change
  2. The intensity of pain when starting the dressing change (remove gauze)
  3. The intensity of pain when at the dressing change (washing the wound)
  4. The intensity of pain when at the end of the dressing change (the dressing is wrapped)
  5. The intensity of pain 30 minutes after the dressing change
Burns Specific Pain Anxiety Scale (BSPAS) : 0 represents not anxious, and 10 represents very anxious | one year
  1. The intensity of anxiety 30 minutes before the dressing change
  2. The intensity of anxiety 30 minutes after the dressing change

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Man Pan, Study Chair — Ditmanson Medical Foundation Chia-Yi Christian Hospital